CLINICAL TRIAL: NCT00858520
Title: Serum, Plasma, DNA and Tissue Bank of Patients With Chronic Obstructive Pulmonary Disease, Lung Cancer and Smoking Controls.
Brief Title: Serum, Plasma, DNA and Tissue Bank in Chronic Obstructive Pulmonary Disease and Lung Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Marc Decramer, Prof.Dr., KU Leuven
Other Study IDs: B32220072389; S50623
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: Chronic Obstructive Pulmonary Disease; Lung Cancer
Keywords: COPD; Lung cancer; genes; DNA
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Germline DNA, serum and plasma, Peripheral blood mononuclear cells, Lung tissue biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Smoking controls: Smokers without lung cancer and without COPD
- COPD patients: Smokers with COPD but without lung cancer
- Lung cancer patients: smokers - never smokers with lung cancer

SUMMARY:
A biobank of Serum, plasma, DNA samples together with clinical information including specific questionnaires, complete pulmonary function and chest CT-scan, is prospectively collected in patients seen at the investigators' clinical service.

The objective is to study candidate gene pathways in COPD and or lung cancer and to associate them with the clinical characteristics and phenotypes of COPD/emphysema and lung cancer.

In subgroups of well characterised patients, other biological materials are also collected (lung tissue biopsies, peripheral blood mononuclear cells).

DETAILED DESCRIPTION:
All patients with a smoking history of at least 15 pack years, an minimal age of 50 years and an recent available CT scan are enrolled.

All subjects with a diagnosis of lung cancer are also collected (irrespective of age and smoking behavior).

In addition the investigators collect:

* specific questionnaires (MRC, CCQ and smoking history)
* medical and professional history
* complete pulmonary function (spirometry, bodyplethysmography and diffusing capacity)
* serum, plasma and DNA samples.

In specific subgroups the investigators also collect:

* Peripheral blood mononuclear cells
* Lung tissue - if available - from a surgical procedure (lung transplantation or lobectomy)

ELIGIBILITY:
Inclusion Criteria for smokers:

* A smoking history of at least 15 pack years and age of 50 years or older
* Complete pulmonary function on day of visit
* Chest CT-scan within one year of enrollment
* 4 weeks from exacerbation

Exclusion Criteria for smokers:

* Less than 15 pack years
* Younger than 50 year
* Other pulmonary diseases interfering with CT or pulmonary function
* Asthma

Inclusion Criteria for lung cancer patients:

* new diagnosis of proven lung cancer
* chest CT scan within 2 months of enrollment
* Complete pulmonary function

Exclusion Criteria for lung cancer patients

* not able to perform pulmonary function
* Absence of histological diagnosis of lung cancer

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Chronic Obstructive Pulmonary Disease and smoking controls.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2007-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Serological, cytological, histological and genetic analysis of biomarkers or genes which are involved in the pathogenesis of COPD/Emphysema/Lungcancer. | 0-1-3-6 years
  All cases are prospectively collected in University hospital Leuven, Belgium. Of enrolled subjects data are collected at 0,1,3 and 6 years interval

CONTACTS AND LOCATIONS:
Overall Officials: Wim Janssens, MD. PhD., Principal Investigator — KU Leuven
Locations (1):
- Katholieke Universiteit Leuven, Leuven, Flanders, Belgium